CLINICAL TRIAL: NCT05684822
Title: The Effects of Acupuncture on Insomnia Among Midlife Women: A Randomized Clinical Trail
Brief Title: The Effects of Acupuncture on Insomnia Among Midlife Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190101
Record Dates: First submitted 2022-10-14; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-10

CONDITIONS: Menopause Syndrome
Keywords: Midlife Women; Acupuncture; Insomnia; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study is designed according to the Impaired Sleep Model, and is a single-blind randomized clinical trial.
Who Masked: Participant
Masking Description: The patients will not know that they are recieving acupuncture or sham acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group received acupuncture treatment (Experimental): The experimental group received acupuncture treatment (Taichong, Shenmen, Neiguan points) twice a week, total three weeks, plus sleep hygiene guidance
  Interventions: Other: Acupuncture
- The control group received subcutaneous sham acupuncture (Sham Comparator): The control group received subcutaneous acupuncture (non-therapeutic acupuncture points) twice a week, total three weeks and given sleep Health guidance.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupoint:Taichong, Shenmen, Neiguan points with twice a week for total three weeks

SUMMARY:
Aims: To explore the effects of acupuncture on the improvement of insomnia, fatigue, depression and menopausal symptoms among midlife women.

DETAILED DESCRIPTION:
This research is a study with a randomized clinical trial. Participants were 40-60 years old with a sleep disturbance which persists more than one month. Twenty participants were randomly assigned into the experimental and control groups. The experimental group received acupuncture treatment (Taichong, Shenmen, Neiguan points) twice a week, total three weeks, plus sleep hygiene guidance; the control group received subcutaneous acupuncture (non-therapeutic acupuncture points) twice a week, total three weeks and given sleep Health guidance. All participants received pre-test and post-test, including sleep multiple physiological examination (PSG), Pittsburgh sleep quality table, Epworth sleepiness scale, hospital anxiety depression scale, menopausal symptom questionnaire, sleep disturbance comprehensive scale, and wore Actiwatch for three days. Data analysis was performed using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-60 years
* Complaints of insomnia symptoms in the past month that lasted for at least one week, such as difficulty falling asleep, waking up easily in the middle of the night, unable to fall asleep after waking up, still not getting enough sleep after waking up in the morning
* The score of sleep disorder on the Pittsburgh Sleep Quality Scale was more than 5 points

Exclusion Criteria:

* History of psychiatric disorders
* History of sleep apnea or nocturnal myoclonus
* Center or neurodegenerative disease
* Cancer
* Melatonin or sleeping pills use in the past month

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 15 minutes
  The scale is suitable for the evaluation of sleep quality in patients with sleep disorders and mental disorders, as well as for the evaluation of sleep quality in general people.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic.
Epworth Sleepiness Scale (ESS) | 15 minutes
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.
Snore Outcomes Survey (SOS) | 15 minutes
  The SOS consists of 8 items relating to the intensity, duration, frequency, and impact of SDB symptoms - specifi cally snoring.
Global Physical Activity Questionnaire | 15 minutes
  The Global Physical Activity Questionnaire was developed by WHO for physical activity surveillance in countries. It collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour, comprising 16 questions (P1-P16)
Total sleep time (TST) | 8 hours
  TST was determined as the number of minutes asleep in bed after "lights off," considering only nighttime sleep.
Wake time after sleep onset (WASO) | 8 hours
  Wake time after sleep onset is time during which one is awake.
Sleep Latency | 8 hours
  Sleep latency, or sleep onset latency, is the time it takes a person to fall asleep after turning the lights out.
Percentage of rapid eye movement (REM) stage | 8 hours
  REM sleep is the stage in which most people vividly dream. These periods of sleep typically start around 90 minutes after someone falls asleep.
Sleep efficiency (SE) | 8 hours
  Sleep efficiency (SE), commonly defined as the ratio of total sleep time (TST) to time in bed (TIB), plays a central role in insomnia research and practice. The significance of SE is understandable because it captures a core problem for those suffering from insomnia-spending too much time in bed trying to sleep.
Minimum spo2 level during sleep | 8 hours
  A normal level of oxygen is usually 95% or higher. Some people with chronic lung disease or sleep apnea can have normal levels around 90%.
Mean heart rate during REM | 8 hours
  Rapid eye movement (REM) sleep is characterized by periods of profound cardiac autonomic activation evident in heart rate surges in humans and canines.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health and Welfare Tainan Hospital, Tainan, Taiwan